CLINICAL TRIAL: NCT06056986
Title: Prospective Study to Evaluate the Role of Shear-Wave Elastography in Predicting the Degree of Intestinal Fibrosis in Patients With Crohn's Disease Who Are Candidates for Surgery - ElChir Study
Brief Title: Shear-Wave Elastography in Intestinal Fibrosis Evaluation in Crohn's Disease
Acronym: EL-CHIR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Zocco Maria Assunta, Prof, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3310
Record Dates: First submitted 2023-03-16; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): Chron's disease patients scheduled for ileo-colonic resection
  Interventions: Diagnostic Test: multimodal ultrasound

INTERVENTIONS:
Diagnostic Test: multimodal ultrasound — Dynamic contrast-enhanced ultrasound and shear wave elastography are perfomed on target intestinal loop

SUMMARY:
The choice of the optimal timing for surgery in Crohn's disease is a challenging issue and diagnostic tools able to estimate the degree of fibrosis are of great interest in this context. Indeed, inflammatory intestinal loops are more likely to respond to medical therapies, wheareas fibrotic loops need to be treated surgically. Shear-wave elastography, which is a non-invasive and largely available technique for the study of tissue elasticity, is very promising and a recent meta-analysis has evaluated its diagnostic accuracy vs histologic examination in patients with stenosing Crohn's disease, showing encouraging results.

Aim of this study is to evaluate the diagnostic agreement between elastographic parameters (mean, median, stability index) and the degree of intestinal fibrosis evaluated on the surgical specimen.

DETAILED DESCRIPTION:
Background: The choice of the optimal timing for surgery in Crohn's disease is a challenging issue and diagnostic tools able to estimate the degree of fibrosis are of great interest in this context. Indeed, inflammatory intestinal loops are more likely to respond to medical therapies, wheareas fibrotic loops need to be treated surgically. Shear-wave elastography, which is a non-invasive and largely available technique for the study of tissue elasticity, is very promising and a recent meta-analysis has evaluated its diagnostic accuracy vs histologic examination in patients with stenosing Crohn's disease, showing encouraging results.

Primary aim: to evaluate the diagnostic agreement between elastographic parameters (mean, median, stability index) and the degree of intestinal fibrosis evaluated on the surgical specimen.

Secondary aims:

* To evaluate the relationship between clinical disease activity assessed by the Harvey Bradshaw index and elastographic parameters.
* To evaluate the concordance between three different methods of shear wave elastography (point and 2D) and different machines.
* To identify elastographic cut-offs capable of predicting the presence and degree of fibrosis.
* To evaluate the agreement between elastography and magnetic resonance imaging (MRI) parameters of fibrosis in a subgroup of patients who underwent MRI preoperatively.

Exploratory aims:

* To evaluate the relationship between elastographic parameters/fibrosis histological score and serum fibrosis biomarkers.
* To evaluate the relationship between elastographic parameters/fibrosis histological score and fecal microbiota.
* To evaluate the changes in serum biomarkers of fibrosis assayed pre- and post-operatively.
* To evaluate the changes in fecal microbiota analyzed pre-and post-operatively Study design: Prospective, interventional, single-center study Methods: Consecutive patients with ileal or ileo-colonic Crohn's disease needing to undergo ileo-cecal resection as per clinical practice with an affected intestinal segment detectable in B-mode ultrasound will be enrolled in the Unit of Internal Medicine and Gastroenterology of the Policlinico Gemelli. Exclusion criteria will be diagnosis of IBD other than Crohn's disease, Crohn's disease without ileal involment, lack of visualization of affected intestinal tract (eg. obesity), hearth failure, known allergy to ultrasound contrast agents, pregnancy and lactation. Considering that the primary objective is the evaluation of the agreement between the parameters obtained from three different elastography and the degree of intestinal fibrosis evaluated on the surgical specimen (histological) and assuming that the disagreement rate (for each single comparison) is 5%, with a confidence level of 0.05 and a power of 80%, a sample size of N=18 subjects is proposed. Upon informed consent, personal data and anamnesis will be collected within 30 days from the scheduled date for surgery (T0) and a venipuncture will be carried out as per normal clinical practice. Subsequently we will proceed with the ultrasound evaluation in B-mode for the identification of the target loop and the elastographic examination with two different ultrasounds (Esaote - MyLabTM9 and Aixplorer Mach 30® - SuperSonic Imagine) and three different technologies (point and 2D Esaote QElaxto ® and ShearWave™ Elastography-Supersonic Imagine). After surgical intervention, fibrosis scores will be calculated on the target loop by an expert Anatomo-Pathologist. Blood tests, ultrasound evaluations (B-mode ultrasound, elastography), surgery and histological examination of the intestinal specimen will be performed as per normal clinical practice. Data obtained from these procedures will be recorded and analyzed specifically for the study. The only study-specific procedures are the collection of fecal samples for microbiota evaluation, urine samples for metabolomics evaluation and an additional blood sample for evaluation of fibrosis biomarkers, all collected at T0 and 6-8 weeks after surgery (T1). The additional blood sample will be taken from the same peripheral venous access route used for blood sampling in normal clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of ileal or ileo-colonic Crohn's disease
* patients scheduled for elective intestinal resection for Crohn's disease within 30 days from enrollment
* affected intestinal segment detectable in B-mode ultrasound

Exclusion Criteria:

* diagnosis of IBD other than Crohn's disease
* Crohn's disease without ileal involment
* lack of visualization of affected intestinal tract (eg. obesity)
* hearth failure
* known allergy to ultrasound contrast agents
* pregnancy
* lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-06-18 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
liver stiffness values useful for assessing intestinal fibrosis and inflammation | 3 months after surgery
  to identify liver stiffness values (kPa) measured with shear-wave elastography that may predict the degree of bowel wall fibrosis or inflammation

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Roma, Italy